CLINICAL TRIAL: NCT00183027
Title: Dietary Energy Restriction and Metabolic Aging in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG0044; 3U01AG020480 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-11-09 (Estimated); Status verified 2006-11

CONDITIONS: Obesity
Keywords: Dietary restriction; Caloric restriction
MeSH Terms: conditions — Obesity | interventions — Energy Intake

INTERVENTIONS:
Behavioral: Dietary composition and energy intake

SUMMARY:
The purpose of this study is to develop an effective calorie restricted diet.

DETAILED DESCRIPTION:
This study is a 3-phase investigation designed to test two caloric restriction (CR) regimens for participant compliance and variability in metabolic and physiologic effects. Initially, and through phase 1 (1 week pre-phase, and 6 weeks phase 1), participants will maintain normal habits at home.

Then for phase 2 (24 weeks), the 44 participants will be randomized to one of two diets (Diet HG or Diet LG), which they will consume at either 70% or 90% of baseline energy intake. The participants randomized to 90% CR (both diets) will form the control group. All food will be provided during this phase, and participants will be required to attend weekly group or individual meetings with the behavioral counselor and dietitian, and perform regular self-monitoring.

During phase 3 (24 weeks), participants will prepare their own food at home according to their CR regimen and will eat to maintain the CR specified for phase 2. They will continue to attend the weekly meetings and to perform self-monitoring.

Diet HG: a diet based on the USDA Food Guide Pyramid, but with additional emphasis on adequate fiber and low energy density foods, including use of whole grains rather than refined carbohydrates, limited liquid calories, high variety of low energy items such as fruits and vegetables and low variety of high-energy discretionary foods.

Diet LG: a modification of the HG diet in which low energy density is maintained even though the percent of energy from fat and protein is increased (by increased use of high-protein foods and foods with high water content) and use of different carbohydrate sources and physically intact food items (whole grains, raw fruits and vegetables) to further lower glycemic load through reducing the glycemic index (GI). High fiber intakes, low energy density, limited use of liquid calories, high variety of low energy items such as fruits and vegetables and low variety of high-energy discretionary foods will be the same as for the HG diet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women (based on standard laboratory tests and a screening examination)
* 20-42 years of age
* BMI in the range 25-29.9 kg/m2
* Proportional representation of minorities in the Greater Boston Area (7 percent Black, 11 percent Hispanic, 82 percent non-Hispanic white)
* Able to accurately complete a food record
* Stage of change >1 for weight loss and changing dietary intake
* Must have an immediate adult family member who is supportive of weight loss

Exclusion Criteria:

* Known serious disorders that affect longevity, energy metabolism, body composition and immune responsiveness, including diabetes, cancer, heart disease, cachexia, eating disorders (anorexia and bulimia and any vomiting for means of weight control), depression, alcoholism, inflammatory disorders and AIDS, and individuals taking medicine that is anticipated to influence lifespan or energy metabolism
* Abnormal kidney function as assessed by serum creatinine, BUN and urinalysis, and abnormal liver function as assessed by SGPT, SGOT alkaline phosphatase, and bilirubin, abnormal normal thyroid function as assessed by serum T4 and TSH and fasting serum glucose levels <125 mg/dl
* Smoking, highly restrained eating, reported endurance training (participation in sports or training >12 hours per week), alcohol intake of 14 oz. per week or more, major medical and/or psychiatric disorders, plans to have a child within 3 years (1 year for Pilot study), past childbearing (for women) within the last 2 years, or breastfeeding within the past year
* Amputees
* Have required treatment for any psychiatric disorder
* Gained or lost >15 lb weight within the past year, or taking medications known or suspected to have an important influence on lifespan, energy metabolism, body composition or immune function
* Early death from cardiovascular diseases, cancer, or a diabetes-related illness (before the age of 45 years) in one or both of the parents
* Unable to remain in the program for at least 1 year, or unsuitable for home-based programs (including individuals reporting binge eating disorders or clinical depression, and women intending to become pregnant)

Ages: 20 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44
Dates: Start 2002-11; Study Completion 2004-12

PRIMARY OUTCOMES:
Changes in body weight, body fatness and total energy expenditure at baseline, 3, 6, and 12 months of caloric restriction (CR).

SECONDARY OUTCOMES:
Changes in blood pressure, insulin sensitivity and secretion, resting metabolic rate, bone mineral density, disease incidence, cognitive function, immune function, oxidative stress parameters, fertility hormones at baseline, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan B. Roberts, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hadley EC, Dutta C, Finkelstein J, Harris TB, Lane MA, Roth GS, Sherman SS, Starke-Reed PE. Human implications of caloric restriction's effects on aging in laboratory animals: an overview of opportunities for research. J Gerontol A Biol Sci Med Sci. 2001 Mar;56 Spec No 1:5-6. doi: 10.1093/gerona/56.suppl_1.5. No abstract available. PMID 12088212
- [Background] Lee IM, Blair SN, Allison DB, Folsom AR, Harris TB, Manson JE, Wing RR. Epidemiologic data on the relationships of caloric intake, energy balance, and weight gain over the life span with longevity and morbidity. J Gerontol A Biol Sci Med Sci. 2001 Mar;56 Spec No 1:7-19. doi: 10.1093/gerona/56.suppl_1.7. PMID 12088215
- [Background] Weindruch R, Keenan KP, Carney JM, Fernandes G, Feuers RJ, Floyd RA, Halter JB, Ramsey JJ, Richardson A, Roth GS, Spindler SR. Caloric restriction mimetics: metabolic interventions. J Gerontol A Biol Sci Med Sci. 2001 Mar;56 Spec No 1:20-33. doi: 10.1093/gerona/56.suppl_1.20. PMID 12088209
- [Background] Mobbs CV, Bray GA, Atkinson RL, Bartke A, Finch CE, Maratos-Flier E, Crawley JN, Nelson JF. Neuroendocrine and pharmacological manipulations to assess how caloric restriction increases life span. J Gerontol A Biol Sci Med Sci. 2001 Mar;56 Spec No 1:34-44. doi: 10.1093/gerona/56.suppl_1.34. PMID 12088210
- [Background] Poehlman ET, Turturro A, Bodkin N, Cefalu W, Heymsfield S, Holloszy J, Kemnitz J. Caloric restriction mimetics: physical activity and body composition changes. J Gerontol A Biol Sci Med Sci. 2001 Mar;56 Spec No 1:45-54. doi: 10.1093/gerona/56.suppl_1.45. PMID 12088211
- [Background] Allison DB, Miller RA, Austad SN, Bouchard C, Leibel R, Klebanov S, Johnson T, Harrison DE. Genetic variability in responses to caloric restriction in animals and in regulation of metabolism and obesity in humans. J Gerontol A Biol Sci Med Sci. 2001 Mar;56 Spec No 1:55-65. doi: 10.1093/gerona/56.suppl_1.55. PMID 12088213
- [Background] Felson DT, Zhang Y, Hannan MT, Kannel WB, Kiel DP. Alcohol intake and bone mineral density in elderly men and women. The Framingham Study. Am J Epidemiol. 1995 Sep 1;142(5):485-92. doi: 10.1093/oxfordjournals.aje.a117664. PMID 7677127
- [Result] Pittas AG, Das SK, Hajduk CL, Golden J, Saltzman E, Stark PC, Greenberg AS, Roberts SB. A low-glycemic load diet facilitates greater weight loss in overweight adults with high insulin secretion but not in overweight adults with low insulin secretion in the CALERIE Trial. Diabetes Care. 2005 Dec;28(12):2939-41. doi: 10.2337/diacare.28.12.2939. No abstract available. PMID 16306558
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717